CLINICAL TRIAL: NCT00600275
Title: A Phase I/II, Multi-center, Open-label Study of BGT226, Administered Orally in Adult Patients With Advanced Solid Malignancies Including Patients With Advanced Breast Cancer
Brief Title: A Phase I/II Study of BGT226 in Adult Patients With Advanced Solid Malignancies Including Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBGT226A2101
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2012-11

CONDITIONS: Solid Tumors; Breast Cancer; Cowden Syndrome
Keywords: BGT226; Solid tumors; Breast cancer; Cowden Syndrome; Phosphatidylinositol 3'-kinase (PI3K) inhibitor; Advanced solid tumors (including sporadic and Cowden Syndrome) (Phase I part); Advanced breast cancer (including sporadic and Cowden Syndrome) (Phase II part)
MeSH Terms: conditions — Breast Neoplasms; Hamartoma Syndrome, Multiple; Hereditary Sensory and Autonomic Neuropathies | interventions — 8-(6-methoxypyridin-3-yl)-3-methyl-1-(4-piperazin-1-yl-3-trifluoromethylphenyl)-1,3-dihydroimidazo(4,5-c)quinolin-2-one

ARMS (1):
- BGT226 (Experimental)
  Interventions: Drug: BGT226

INTERVENTIONS:
Drug: BGT226

SUMMARY:
This is a phase I/II clinical research study with BGT226, an inhibitor of phosphatidylinositol 3'-kinase (PI3K). The study consists of a Phase I dose escalation part followed by a safety expansion part and a Phase II expansion part.

Once the MTD has been defined, the safety expansion and efficacy expansion parts of the trial will be opened for enrollment.

Phase I safety expansion part will enroll advanced solid tumors. Phase II expansion part will enroll advanced breast cancer. An effort will be made to enrich the trial population with Cowden Syndrome patients with advanced solid malignancies.

ELIGIBILITY:
Inclusion criteria:

All patients

* Histologically-confirmed, advanced solid tumors
* Progressive, recurrent unresectable disease

Phase II expansion part (advanced breast cancer)

* Confirmed positive hormone receptor (estrogen receptor and/or progesterone receptor) or positive HER-2 expression status
* Disease progression/recurrence following hormonal or anti-HER-2 treatment for advanced disease
* At least one but not more than two prior chemotherapy regimens for the unresectable tumor
* Measurable disease by MRI or CT scan

Cowden Syndrome patients with an advanced malignancy Genetic confirmation of Cowden Syndrome

* Age ≥ 18
* World Health Organization (WHO) Performance Status of ≤ 2

Exclusion criteria:

* Hematopoietic:
* No diabetes mellitus or history of gestational diabetes mellitus
* No acute or chronic renal disease
* No acute or chronic liver disease
* No acute or chronic pancreatitis
* No impaired cardiac function or clinically significant cardiac diseases such as ventricular arrhythmia, congestive heart failure, uncontrolled hypertension
* No acute myocardial infarction or unstable angina pectoris within the past 3 months
* Not pregnant or nursing and fertile patients must use barrier contraceptives

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of BGT226 (Phase I dose escalation) Safety and tolerability of BGT226 (all patients) Clinical tumor response in patients with advanced breast cancer (Phase II) | throughout the study

SECONDARY OUTCOMES:
Pharmacodynamics Changes in biological markers indicative of the inhibitory effect of BGT226. Changes in cellular physiology as assessed by Positron Emission Tomography (PET) imaging | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - Nevada Cancer Center, Las Vegas, Nevada
  - Cancer Therapy and Research Center (CTRC), San Antonio, Texas
- Princess Margaret Hospital, Toronto, Canada
- Novartis Investigative Site, Barcelona, Spain

REFERENCES:
- See also: Results for CBGT226A2101 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3640